CLINICAL TRIAL: NCT00672464
Title: Combined Treatment of Cardiovascular Risk Factors In Newly Admitted Patients With Schizophrenia or Schizoaffective Disorder Who Are Receiving Olanzapine And Matched Controls
Brief Title: Cardio Risk of Acute Schizophrenia Olanzapine Duke
Acronym: CRASOD
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: Pro00006916; None (investigator sponsored)
Record Dates: First submitted 2008-05-04; First posted 2008-05-06 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective; Cardiovascular; Olanzapine; Metformin; Simvastatin
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Olanzapine; Metformin; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Olanzapine only (Active Comparator): Newly Admitted Patients with Schizophrenia or Schizoaffective Disorder Who Are Receiving Olanzapine
  Interventions: Drug: Olanzapine
- Added Metformin (Experimental): Newly Admitted Patients with Schizophrenia or Schizoaffective Disorder Who Are Receiving Olanzapine with Added Metformin
  Interventions: Drug: Olanzapine; Drug: Metformin
- Added Simvastatin (Experimental): Newly Admitted Patients with Schizophrenia or Schizoaffective Disorder Who Are Receiving Olanzapine with Added Simvastatin
  Interventions: Drug: Olanzapine; Drug: Simvastatin
- Added Metf. + Simv. (Experimental): Newly Admitted Patients with Schizophrenia or Schizoaffective Disorder Who Are Receiving Olanzapine with Added Metformin and Simvastatin
  Interventions: Drug: Olanzapine; Drug: Metformin; Drug: Simvastatin
- Matched Controls (No Intervention): Matched Control Subjects by age, race, and gender

INTERVENTIONS:
Drug: Olanzapine — Olanzapine zydis 15 mg QHS for 28 days
  Arms: Added Metf. + Simv.; Added Metformin; Added Simvastatin; Olanzapine only
Drug: Metformin — Metformin capsules will be started at 500 mg twice a day (before breakfast and before dinner) for days 1-3, then 500 mg before breakfast and 1000 mg before dinner for days 4-7, and then 1000 mg twice a day thereafter.
  Arms: Added Metf. + Simv.; Added Metformin
Drug: Simvastatin — Simvastatin will be started at 10 mg at bed time for the first week and 20 mg at bedtime thereafter.
  Arms: Added Metf. + Simv.; Added Simvastatin

SUMMARY:
Primary Objective: To compare added metformin and/or added simvastatin versus no intervention in reducing or eliminating increased cardiovascular risk (as estimated by elevation in non-HDL cholesterol levels) during the treatment of schizophrenia with olanzapine.

Secondary Objective(s): To compare added metformin and/or added simvastatin versus no intervention in reducing or eliminating increased cardiovascular risk (as estimated by elevation in triglyceride levels) during the treatment of schizophrenia with olanzapine. To compare added metformin and/or added simvastatin versus no intervention in reducing or eliminating increased cardiovascular risk (as estimated by C-reactive protein levels) during the treatment of schizophrenia with olanzapine

DETAILED DESCRIPTION:
Olanzapine offers greater therapeutic antipsychotic benefit than the other non-clozapine antipsychotic medications available in the U.S., making it a desirable choice for the long-term maintenance treatment of patients with schizophrenia (Lieberman et al, 2005). Long-term compliance with an efficacious antipsychotic medication is fundamental to optimal therapeutic outcomes. Toward this goal, a long-acting injectable preparation of olanzapine will soon be available.

However, the long-term use of olanzapine has been limited by its substantial, un-wanted effects on metabolism that result in weight gain, increases in insulin resistance, increases in non-HDL-cholesterol, and increases in C-reactive protein (Lieberman et al, 2005; McEvoy et al, 2005;Meyer et al, 2008; McEvoy et al, in submission). Over the long term, insulin resistance contributes to the accelerated incidence of diabetes mellitus that has been observed among patients with schizophrenia since the availability of the atypical antipsychotic medication (Basu A, 2006). Over the long term, elevated non-HDL-cholesterol and increased inflammation contribute independently to the accelerated cardiovascular mortality that has been observed among patients with schizophrenia since the availability of the atypical antipsychotic medications (Saha et al, 2007, Capasso et al, 2007). Inflammation, as measured by C-reactive protein, provides added, independent predictive value of cardiovascular risk beyond that of measures of insulin resistance and elevated non-HDL-cholesterol.

Established strategies exist that may attenuate these unwanted effects of olanzapine on metabolism and inflammation. Metformin has been shown to reduce weight gain and insulin resistance in pre-diabetic, obese individuals without mental problems (Salpeper et al, 2008) and in patients treated with atypical antipsychotic medications (Wu et al, 2008). Statins have been shown to reduce non-HDL-cholesterol and cardiovascular morbidity and mortality (Lee et al, 2007). Both metformin and statins have been shown to reduce C-reactive protein (Bulcau et al, 2007).

We propose to implement a pilot study to estimate the effects sizes (for change in triglycerides, change in non-HDL-cholesterol, and change in CRP) of added metformin, added simvastatin, or added metformin and simvastatin, versus added no intervention in 120 newly-admitted, acutely psychotic, recently un-medicated patients with schizophrenia over 4 weeks of prospective treatment with olanzapine. We will also compare these patients (baseline values, in the not recently medicated state) to 40 age, race, and gender matched control subjects on fasting triglycerides, non-HDL-cholesterol, and CRP levels.

We will recruit newly admitted patients experiencing an acute psychotic relapse of schizophrenia (related to failure to take their prescribed antipsychotic medication). After baseline assessments and samplings have been completed, all patient will be treated with olanzapine zydis 15 mg QHS for 28 days. All patients will be randomized 1:1:1:1 to added metformin, added simvastatin, added metformin and simvastatin, or no intervention. All treatments will be open label. Repeated assessments of weight, non-HDL-cholesterol, triglycerides and C-reactive protein will be obtained. Subjects will remain as inpatients at JUH for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* We will include patients who come to us free of antipsychotic medication, i.e., patients with chronic schizophrenia (with at least one prior psychiatric hospitalization) who have been off antipsychotic medication for at least 3 weeks and who are newly hospitalized for treatment of an acute psychotic relapse; these patients will be male or female, 18-60 years of age, meet DSM-IV criteria for schizophrenia, and have scores >=4 on at least two of the PANSS Positive subscale items.

Exclusion Criteria:

* We will exclude patients whose psychoses are predominantly affective in nature or explainable on the basis of substance abuse or a co-morbid medical condition, patients with diabetes mellitus, epilepsy, mental retardation, or organic mental syndromes, and patients currently taking metformin or a statin.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2009-12 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
To compare added metformin and/or added simvastatin versus no intervention in reducing or eliminating increased cardiovascular risk (as estimated by elevation in non-HDL cholesterol levels) during the treatment of schizophrenia with olanzapine. | 28 days

SECONDARY OUTCOMES:
To compare added metformin and/or added simvastatin versus no intervention in reducing or eliminating increased cardiovascular risk during the treatment of schizophrenia with olanzapine. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P McEvoy, MD, Principal Investigator — Duke University Medical Center, Dep't. Psychiatry
Locations (2):
- United States (2):
  - John Umstead Hospital, Butner, North Carolina
  - Duke University Medical Center, Durham, North Carolina